CLINICAL TRIAL: NCT05531279
Title: A Randomized,Open-label Dose-discovery Study of PEG-rhG-CSF and rhG-CSF in the Adjuvant Therapy of Aplastic Anemia Granulocyte Deficiency
Brief Title: A Study of PEG-rhG-CSF and rhG-CSF Used for Aplastic Anemia Granulocyte Deficiency
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT2021022-EC-1
Record Dates: First submitted 2022-09-02; First posted 2022-09-07 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2022-09

CONDITIONS: Severe Aplastic Anemia
Keywords: G-CSF
MeSH Terms: conditions — Anemia, Aplastic | interventions — pegylated granulocyte colony-stimulating factor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PEG-rhG-CSF group A (Experimental): PEG-rhG-CSF group A(q7d):6mg d1,8,subcutaneously injected,after monitoring ANC>0.5×109/L,the drug was stopped,and then ANC<0.5×109/L was temporarily supplemented with one dose of the same drug.
  Interventions: Drug: PEG-rhG-CSF
- PEG-rhG-CSF group B (Experimental): PEG-rhG-CSF group B(q10d):6mg d1,11,subcutaneously injected,after monitoring ANC>0.5×109/L,the drug was stopped,and then ANC<0.5×109/L was temporarily supplemented with one dose of the same drug.
  Interventions: Drug: PEG-rhG-CSF
- rhG-CSF group(short-acting ) (Experimental): rhG-CSF group(short-acting ): 480ug d1-14(daily for 14days),subcutaneously injected.After monitoring ANC>0.5×109/L,the drug was stopped,and then ANC<0.5×109/L was temporarily supplemented with one dose of the same drug.
  Interventions: Drug: PEG-rhG-CSF

INTERVENTIONS:
Drug: PEG-rhG-CSF — PEG-rhG-CSF group A(q7d):6mg d1,8,subcutaneously injected; PEG-rhG-CSF group B(q10d):6mg d1,11,subcutaneously injected; RhG-CSF group(short-acting ): 480ug d1-14(daily for 14days),subcutaneously injected.
  Other Names: rhG-CSF

SUMMARY:
This study was a single-center,open-label,randomized,dose-exploring prospective study.Patients with granulocytotic aplastic anemia who received cytokine treatment with PEG-rhG-CSF or rhG-CSF were enrolled.Clinical demographic data,disease characteristics of aplastic anemia,clinical diagnosis and treatment,laboratory data and adverse events were collected to explore the dose and safety of PEG-rhG-CSF and rhG-CSF in patients with severe aplastic anemia.

DETAILED DESCRIPTION:
This study was a single-center,open-label,randomized,dose-exploring prospective study.Patients with granulocytotic aplastic anemia who received cytokine treatment with PEG-rhG-CSF or rhG-CSF were enrolled.Clinical demographic data,disease characteristics of aplastic anemia,clinical diagnosis and treatment,laboratory data and adverse events were collected to explore the dose and safety of PEG-rhG-CSF and rhG-CSF in patients with severe aplastic anemia.Research objectives: To explore the reasonable injection frequency of long-acting PEG-rhG-CSF in the adjuvant treatment of aplastic anemia patients with granulocytosis through a single center prospective clinical study.Disease classification of aplastic anemia: a total of 45 cases of SAA/VSAA with ANC<0.5×109/L were stratified and randomized into three groups according to the radio of 1:1:1(15 cases in each group).PEG-rhG-CSF group A(q7d):6mg d1,8,subcutaneously injected;PEG-rhG-CSF group B(q10d):6mg d1,11,subcutaneously injected;RhG-CSF group(short-acting ): 480ug d1-14(daily for 14days),subcutaneously injected.Dose/protocol adjustment: after monitoring ANC>0.5×109/L,the drug was stopped,and then ANC<0.5×109/L was temporarily supplemented with one dose of the original group of drugs.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years old, male or female, or weight≥50kg.
2. Patients with severe or very severe aplastic anemia of absolute neutrophil value< 0.5×109/L
3. ECOG score ≤ 2 points.
4. Normal renal function.

Exclusion Criteria:

1. Patients with clonal chromosomal abnormalities.
2. Patients with previous malignant tumors.
3. Patients with severe or uncontrolled infectious diseases and /or bleeding.
4. Patients with AIDS or syphilis positive.
5. Severe organ dysfunction.
6. Patients used GM/G-CSF,PEG-rhG-CSF,interleukin-11 within 2 weeks before admission.
7. Allergic to G-CSF or PEG-rhG-CSF related components.
8. Participated in other clinical trials within 6 months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2022-06-05 (Actual); Primary Completion 2025-06-05 (Estimated); Study Completion 2026-01-05 (Estimated)

PRIMARY OUTCOMES:
total number of effective (ANC>0.5×109/L) days | 2 weeks
  total number of effective (ANC>0.5×109/L) days during 2 weeks of treatment(cases×days).

CONTACTS AND LOCATIONS:
Overall Officials: Liping Jing, Doctor, Study Director — Chinese Academy of Medical Sciences
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
We can share the plan after completing the experiment
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Follow-up and publication of the paper are planned for December 2025
Access Criteria: After the paper is written and published

REFERENCES:
- [Result] Tichelli A, Schrezenmeier H, Socie G, Marsh J, Bacigalupo A, Duhrsen U, Franzke A, Hallek M, Thiel E, Wilhelm M, Hochsmann B, Barrois A, Champion K, Passweg JR. A randomized controlled study in patients with newly diagnosed severe aplastic anemia receiving antithymocyte globulin (ATG), cyclosporine, with or without G-CSF: a study of the SAA Working Party of the European Group for Blood and Marrow Transplantation. Blood. 2011 Apr 28;117(17):4434-41. doi: 10.1182/blood-2010-08-304071. Epub 2011 Jan 13. PMID 21233311